CLINICAL TRIAL: NCT06967857
Title: Randomized, Placebo-controlled Clinical Trial to Investigate the Safety and Efficacy of Two Dexamfetamine Sulfate Formulations in Adults With ADHD and Moderate to Severe Depression (DEXAD)
Brief Title: Clinical Trial to Investigate the Safety and Efficacy of Two Dexamfetamine Sulfate Formulations in Adults With ADHD and Moderate to Severe Depression
Acronym: DEXAD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Frank Behrens (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Frank Behrens, Deputy Head of Institute, Clinical Professor, Head of Department of Clinical Research at ITMP, Fraunhofer Institute for Translational Medicine and Pharmacology ITMP
Organization: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMP-18122023-58
Record Dates: First submitted 2025-04-22; First posted 2025-05-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD); Depression - Major Depressive Disorder
Keywords: ADHD; Depression; Adults
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Depression

STUDY DESIGN:
Intervention Model Description: randomised, double blind
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DEX IR (Experimental): tablets twice daily
  Interventions: Drug: DEX IR tablets
- DEX XL (Experimental): capsule once daily
  Interventions: Drug: DEX XL
- PLC (Placebo Comparator): tablet or capsule as comparator to verum
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DEX IR tablets — tablet twice daily
  Arms: DEX IR
Drug: DEX XL — capsule once daily
  Arms: DEX XL
Drug: Placebo — Placebo to either capsule or tablet
  Arms: PLC

SUMMARY:
The indication of attention-deficit/hyperactivity disorder (ADHD) to be examined often occurs with other psychiatric disorders, and the majority of adults with ADHD have at least one psychiatric comorbidity in their lives. Depression is one of the most common comorbidities in patients with ADHD. The prevalence of comorbid depression in adults with ADHD is estimated to be as high as 50%.

There is evidence that stimulants such as dexamfetamine and methylphenidate lead to an improvement in sustained focused attention, working memory, and a variety of cognitive processes in the prefrontal cortex (PFC). In combination with the pharmacological effects of stimulants, such as the inhibition of monoamine oxidase, the increase in the concentration of noradrenaline in the PFC and dopamine in the striatum, dexamfetamine and methylphenidate could improve the treatment of depression in patients with major depressive disorder and comorbid ADHD.

This clinical trial will evaluate the safety and efficacy of DEX in two different formulations compared to placebo in adults with ADHD and moderate to severe depression. To ensure double blinding of the treatment, placebo will be administered in the form of tablets and capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of attention deficit / hyperactivity disorder (ADHD) (according to DSM-5 (fifth version of Diagnostic and Statistical Manual of Mental Disorders) or ICD (International Statistical Classification Of Diseases And Related Health Problems) guidelines) which started in childhood (at the age of <12 years)
2. Patient has a minimum ADHS-Diagnostische Checkliste-Q (ADHS-DC) total score of 32 at baseline (Visit (V) 0)
3. Moderate to severe depression according to ICD-10 (depressive episode: Code F32; recurrent depressive disorder: Code F33) and with a Montgomery-Åsberg Depression Rating Scale (MADRS) score of >20 at baseline (V0)
4. CGI-S ≥ 4 at baseline (V0)
5. Patients receiving selective serotonin reuptake inhibitors (SSRIs) or Serotonin-norepinephrine reuptake inhibitors (SNRIs) (stable doses within the last 2 weeks before inclusion) (≤40 mg (es)citalopram, 50-200 mg sertraline, 75 - 300 mg venlafaxine extended release)
6. Male or female patients ≥ 18 years and ≤ 65 at time of enrolment
7. Patients with QTc interval within normal ranges (≤470 ms in males and ≤480 ms in females)
8. Patient is either free of stimulant medication or who, after discussion with his / her treating physician, is able and willing to discontinue the current psychotropic medication(s) for treatment of ADHD symptoms (specifically, methylphenidate, lisdexamfetamine, guanfacine or atomoxetine or any other medication approved for the treatment of ADHD) ) for the duration of the study, as well as is able and willing to discontinue all relevant co-medication according to exclusion criterion no. 20a-s for comorbid conditions during the clinical trial, if applicable
9. Written informed consent and data protection declaration obtained prior to the initiation of any protocol required procedures
10. Willing and able to comply to study procedures and study protocol

Exclusion Criteria:

1. Current or a history of severe co-morbid symptoms such as psychotic symptoms, schizophrenia, bipolar disorders or manic episodes
2. Current or recent history of substance abuse disorder within the last 6 months of clinical trial entry
3. Patients with body mass index (BMI) < 18.5 kg/m² or >35 kg/m²
4. History of serotonin syndrome events
5. History of seizures or use of anticonvulsant medication
6. Any other uncontrolled psychiatric condition that requires medication or may interfere with trial participation
7. Known symptomatic cardiovascular disease including structural abnormalities, moderate and severe hypertension (systolic blood pressure ≥160 mmHg, diastolic blood pressure ≥100 mmHg), heart failure, myocardial infarction, arterial occlusive disease, angina, haemodynamically significant congenital heart disease, cardiomyopathies, potentially life-threatening arrhythmias and channelopathies (diseases caused by ion channel dysfunction)
8. Significant, in the discretion of the investigator, hepatic, gastrointestinal, renal, haematological or oncologic disorder
9. Diagnosis of glaucoma, hyperthyroidism, pheochromocytoma or porphyria
10. Diagnosis or family history of Tourette's syndrome or dystonia
11. Pre-existing cerebrovascular disorders such as cerebral aneurysm, vascular abnormalities including vasculitis or stroke
12. Immunodeficiency disorders (e.g. organ transplantation, Human Immunodeficiency Virus (HIV) infection)
13. Known hypersensitivity to any of the ingredients of the trial medication, e.g. patients with known rare hereditary problems of fructose intolerance
14. Males or females of reproductive potential not willing to use effective contraception (defined as PEARL index <1 - e.g. contraceptive pill, intrauterine device (IUD)) during the study period (Screening to Follow-up)
15. Pregnancy and lactation
16. Participation in another interventional clinical trial during the trial and within the previous 30 days prior to trial start
17. Patients who are institutionalised by court order or regulatory action
18. Patients, who are members of the staff of the trial centre, staff of the sponsor or involved Clinical Research Organisation (CRO), the investigator him- / herself or close relatives of the investigator
19. Legal incapacity and/ or other circumstances rendering the patient unable to understand the nature, scope and possible impact of the clinical trial
20. Current use of and use within the last 2 weeks before inclusion due to possible interactions with stimulants or SSRIs/SNRIs and possible resulting or expected side effects:

    1. Antipsychotics (such as chlorpromazine, haloperidol, thioridazine; except for quetiapine up to 100mg/day)
    2. SSRIs and SNRIs daily doses of >40 mg (es)citalopram, >200 mg sertraline, >300 mg venlafaxine extended release
    3. Monoamine oxidase inhibitors (MAO) inhibitors
    4. tricyclic antidepressants
    5. benzodiazepines (including Z-drugs)
    6. atypical antidepressants (with an exception for daily doses of 100-300 mg trazodone)
    7. Dopamine reuptake inhibitors (special restriction for bupropion)
    8. antiarrhythmics (Class IA and III)
    9. antibiotics (in particular macrolides and fluoroquinolones, linezolid)
    10. opioids
    11. hydroxychloroquine, chloroquine
    12. ketoconazole
    13. acetylsalicylic acid (dose up to 300 mg allowed)
    14. diphenhydramine
    15. apixaban
    16. metoprolol
    17. pregabalin
    18. budesonide / formoterol
    19. albuterol / salbutamol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) in the active treatment groups compared to the placebo until V6 | from enrollment to the end of study at week 17
  Incidence of adverse events (AE) in the active treatment groups (DEX XL and DEX IR) compared to the placebo until V6

SECONDARY OUTCOMES:
Incidence of adverse events (AE) until V5 | Start with enrollment until end of treatment at Week 16
  Dokumentation of AE
Proportion of patients with at least one AE until V5 | through study treatment (up to 16 weeks)
  Proportion of patients with at least one AE until V5
Proportion of patients with at least one AE until end of study | from baseline until end of study at week 17
  Proportion of patients with at least one AE until end of study
Number of AE until V5 | through study treatment (up to 16 weeks)
  Number of AE
Number of AE until V5 and until end of study | from baseline until end of study at week 17
  Number of AE
Number of AE/SAE during the study period | through study treatment (up to 16 weeks)
  Number of AE/SAE
number of patients with AE/SAE by type during study period | through study treatment (up to 16 weeks)
  Number and type of AE/SAE
proportion of patients with AE/SAE by type during study period | through study treatment (up to 16 weeks)
  Proportion of patient with AE/SAE by type
number of patients with AE/SAE by severity (mild, moderate, severe) during study period | through study treatment (up to 16 weeks)
  number of patients with AE/SAE by severity (mild, moderate, severe)
proportion of patients with AE/SAE by severity (mild, moderate, severe) during study period | through study treatment (up to 16 weeks)
  proportion of patients with AE/SAE by severity (mild, moderate, severe)
number of patients with AE/SAE by relatedness to treatment during study period | through study treatment (up to 16 weeks)
  number of patients with AE/SAE by relatedness to treament
proportion of patients with AE/SAE by relatedness to treatment during study period | from enrollment to the end of study at week 17
  proportion of patients with AE/SAE by relatedness to treatment
Score of clinical global impression (CGI) Efficacy index by investigator at Visit 5 | 16 weeks after treatment start
  Clinical global impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in patients with mental disorders. It is a brief 3-item observer-rated scale. 4×4 rating scale that assesses the therapeutic effect of treatment with psychiatric medication and associated side effects. Treatment is evaluated from "marked improvement" to "none/worsening". Side effects is evaluated from "none" to "outweigh therapeutic effect"
MADRS suicidal ideation score for all available visits (screening to Visit 5) | from enrollment to the end of treatment (up to week 16)
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
MADRS suicidal ideation score for all available visits | from enrollment to end of titration at week 4 (V1)
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
MADRS suicidal ideation score for all available visits | from enrollment to week 7 (V2)
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
MADRS suicidal ideation score change to BL/V0 (on V1) | from baseline to end of treatment titration phase at 4 weeks
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
MADRS suicidal ideation score change to BL/V0 (on V5) | from treatment start to end of treatment at 16 weeks
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
MADRS suicidal ideation score for all available visits | from enrollment to 10 weeks (V3)
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
MADRS suicidal ideation score for all available visits | from enrollment to 13 weeks (V4)
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
MADRS suicidal ideation score for all available visits (screening to visit 5) | from enrollment to 16 weeks (V5)
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
Rate of patients with score 1-3 in CGI-I at V5 | from baseline to 16 weeks (V5)
  The clinical global impression - improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Clinicians ask: "Compared to the patient's condition at baseline, this patient's [average] condition has...?" and rated as:
  Very much improved Much improved Minimally improved No change Minimally worse Much worse Very much worse
Absolute scores categories of CGI-I at all available visits | from end of treatment titration phase at 4 weeks (V1) to week 7 (V2)
  The clinical global impression - improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Clinicians ask: "Compared to the patient's condition at baseline, this patient's [average] condition has...?" and rated as:
  Very much improved Much improved Minimally improved No change Minimally worse Much worse Very much worse
Absolute scores categories of CGI-I at all available visits (V1 to V2) | from end of titration phase (week 4) to 7 weeks (V2)
  The clinical global impression - improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Clinicians ask: "Compared to the patient's condition at baseline, this patient's [average] condition has...?" and rated as:
  Very much improved Much improved Minimally improved No change Minimally worse Much worse Very much worse
Absolute scores categories of CGI-I at all available visits (V1 to V3) | from end of titration phase (week 4) to 10 weeks (V3)
  The clinical global impression - improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Clinicians ask: "Compared to the patient's condition at baseline, this patient's [average] condition has...?" and rated as:
  Very much improved Much improved Minimally improved No change Minimally worse Much worse Very much worse
Absolute scores categories of CGI-I at all available visits (V1 to V4) | from end of titration phase (week 4) to 13 weeks (V4)
  The clinical global impression - improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Clinicians ask: "Compared to the patient's condition at baseline, this patient's [average] condition has...?" and rated as:
  Very much improved Much improved Minimally improved No change Minimally worse Much worse Very much worse
Absolute scores categories of CGI-I at all available visits (V1 to V5) | from end of titration phase (week 4) to end of treatment at 16 weeks (V5)
  The clinical global impression - improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Clinicians ask: "Compared to the patient's condition at baseline, this patient's [average] condition has...?" and rated as:
  Very much improved Much improved Minimally improved No change Minimally worse Much worse Very much worse
Numbers and percentages of patients with (1) decreased, (2) maintained and (3) increased CGI-S at V5 compared to BL/V0 | from baseline to end of treatment at 16 weeks (V5)
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Clinicians ask: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" Possible ratings are:
  Normal, not at all ill Borderline mentally ill Mildly ill Moderately ill Markedly ill Severely ill Among the most extremely ill patients
Shift table of CGI-S score categories at BL/V0 | at baseline
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Clinicians ask: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" Possible ratings are:
  Normal, not at all ill Borderline mentally ill Mildly ill Moderately ill Markedly ill Severely ill Among the most extremely ill patients
Shift table of CGI-S score categories at V1 | from baseline to end of treatment titration phase at 4 weeks (V1)
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Clinicians ask: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" Possible ratings are:
  Normal, not at all ill Borderline mentally ill Mildly ill Moderately ill Markedly ill Severely ill Among the most extremely ill patients
Shift table of CGI-S score categories at V5 | from baseline to end of treatment at 16 weeks (V5)
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Clinicians ask: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" Possible ratings are:
  Normal, not at all ill Borderline mentally ill Mildly ill Moderately ill Markedly ill Severely ill Among the most extremely ill patients
Absolute score categories of CGI-S at V0 | at baseline (V0)
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Clinicians ask: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" Possible ratings are:
  Normal, not at all ill Borderline mentally ill Mildly ill Moderately ill Markedly ill Severely ill Among the most extremely ill patients
Absolute score categories of CGI-S at V0 to V2 | from baseline to 7 weeks (V2)
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Clinicians ask: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" Possible ratings are:
  Normal, not at all ill Borderline mentally ill Mildly ill Moderately ill Markedly ill Severely ill Among the most extremely ill patients
Absolute score categories of CGI-S at V0 to V1 | from baseline to end of treatment titration phase at 4 weeks (V1)
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Clinicians ask: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" Possible ratings are:
  Normal, not at all ill Borderline mentally ill Mildly ill Moderately ill Markedly ill Severely ill Among the most extremely ill patients
Absolute score categories of CGI-S at V0 to V3 | from baseline to 10 weeks (V3)
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Clinicians ask: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" Possible ratings are:
  Normal, not at all ill Borderline mentally ill Mildly ill Moderately ill Markedly ill Severely ill Among the most extremely ill patients
Absolute score categories of CGI-S at V0 to V4 | from baseline to 13 weeks (V4)
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Clinicians ask: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" Possible ratings are:
  Normal, not at all ill Borderline mentally ill Mildly ill Moderately ill Markedly ill Severely ill Among the most extremely ill patients
Absolute score categories of CGI-S at V0 to V5 | from baseline to end of treatment at 16 weeks (V5)
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Clinicians ask: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" Possible ratings are:
  Normal, not at all ill Borderline mentally ill Mildly ill Moderately ill Markedly ill Severely ill Among the most extremely ill patients
MADRS total score (range 0-60) for all available visits (SCR to V5) | Screening until end of treatment at week 16 (V5)
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
MADRS total score (range 0-60) MADRS total score (range 0-60) change to BL/V0 (at V5) | baseline until end of treatment at week 16 (V5)
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
MADRS total score categorization by Müller et al. at BL/ V0 | at baseline
  MADRS total score categorization by Müller et al.: 0-6 absence of symptoms; 7-19 mild depression, 20-34 moderate depression, 35-60 indicate a severe depression.
ADHS-DC-Q total score (range 0-66) for all available visits (SCR to V5) | Screening to end of treatment at week 16
  The ADHS-DC-Q consists of 18 items with a four-level response (not existing, slightly existing, moderately existing, strongly existing). The items ask about the current symptoms. The three scales are: lack of inattentiveness, hyperactivity and impulsiveness.
ADHS-DC-Q total score (range 0-66) change to BL/V0 (V1) | from baseline to end of titration at week 4 (V1)
  The ADHS-DC-Q consists of 18 items with a four-level response (not existing, slightly existing, moderately existing, strongly existing). The items ask about the current symptoms. The three scales are: lack of inattentiveness, hyperactivity and impulsiveness.
QIDS-SR-16 total score (range 0-27) for all available visits (V0 to V5) | baseline to end of treatment at 16 weeks
  QIDS-SR-16 is a self-report measure of depression consisting of 16 items. Questions in the QIDS - SR-16 correlate with the nine DSM-IV symptom criterion domains, Including: Sleep disturbance (initial, middle, and late insomnia or hypersomnia), Sad mood, Decrease/increase in appetite/weight , Concentration , Self-criticism, Suicidal ideation, Interest, Energy/fatigue, Psychomotor agitation/retardation. Scoring is given from 0 to 3 whereas 0 indicates less impact, 3 highest impact in depression.
QIDS-SR-16 total score (range 0-27) change to BL/V0 (V5) | from baseline to end of treatment at week 16 (V5)
  QIDS-SR-16 is a self-report measure of depression consisting of 16 items. Questions in the QIDS - SR-16 correlate with the nine DSM-IV symptom criterion domains, Including: Sleep disturbance (initial, middle, and late insomnia or hypersomnia), Sad mood, Decrease/increase in appetite/weight , Concentration , Self-criticism, Suicidal ideation, Interest, Energy/fatigue, Psychomotor agitation/retardation. Scoring is given from 0 to 3 whereas 0 indicates less impact, 3 highest impact in depression.
Mean dose intake from V1 to V5 per treatment group | from end of titration (week 4, V1) until end of treatment at week 16
  Mean dose intake from V1 to V5 per treatment group
Mean dose intake compared to planned dose after titration phase (for study period V1 to V5) per treatment group | end of titration phase (visit 1) 4 weeks after baseline until end of treatment at week 16 (12 weeks after titration phase)
  Mean dose intake compared to planned dose after titration phase per treatment group
Proportion of patients with less than 80% of planned dose intake (for study period V1 to V5) per treatment group | visit 1 (4 weeks after baseline) until end of treatment at week 16
  Proportion of patients with less than 80% of planned dose intake per treatment group
Number of patients by dosage group at V1 and V2 | at visit 1 (4 weeks after baseline) and at visit 2 (3 weeks after visit 1)
  Number of patients by dosage group (DEX IR: 10 mg, 15 mg, 20 mg, 30 mg; DEX XL: 10 mg, 15 mg, 20 mg, 30 mg; Placebo: 10 mg, 15 mg, 20 mg, 30 mg))
Proportion of patients by dosage group at V1 and V2 | at visit 1 (4 weeks after baseline) and at visit 2 (3 weeks after visit 1)
  Proportion of patients by dosage group (DEX IR: 10 mg, 15 mg, 20 mg, 30 mg; DEX XL: 10 mg, 15 mg, 20 mg, 30 mg; Placebo: 10 mg, 15 mg, 20 mg, 30 mg))
Number of patients per treatment group that needed dose optimization of IMP in the optimal stable dose phase and type of optimization (e.g., downtitration) | end of titration phase (visit 1) 4 weeks after baseline until end of treatment at week 16 (12 weeks after titration phase)
  Number of patients per treatment group that needed dose optimization of IMP in the optimal stable dose phase and type of optimization (e.g., downtitration)
Proportion of patients per treatment group that needed dose optimization of IMP in the optimal stable dose phase and type of optimization (e.g., downtitration) | end of titration phase (visit 1) 4 weeks after baseline until end of treatment at week 16 (12 weeks after titration phase)
  Proportion of patients per treatment group that needed dose optimization of IMP in the optimal stable dose phase and type of optimization (e.g., downtitration)
Number of patients with early withdrawal from therapy due to adverse events | baseline until end of treatment at week 16 (12 weeks after end of titration phase)
  Number of patients with early withdrawal from therapy due to adverse events in total
Number of patients with early withdrawal from therapy due to adverse events per treatment group | baseline until end of treatment at week 16 (12 weeks after end of titration phase)
  Number of patients with early withdrawal from therapy due to adverse events per treatment group
percentage of patients with early withdrawal from therapy due to adverse events in total | baseline until end of treatment at week 16 (12 weeks after end of titration phase)
  Percentage of patients with early withdrawal from therapy due to adverse events - in total
Percentage of patients with early withdrawal from therapy due to adverse events per treatment group | baseline until end of treatment at week 16 (12 weeks after end of titration phase)
  Percentage of patients with early withdrawal from therapy due to adverse events per treatment group
MADRS total score categorization by Müller et al. at BL/ V0, V1 and V5 | at baseline, at end of titration phase (week 4) and at end of treatment (week 16, V5)
  MADRS total score categorization by Müller et al.: 0-6 absence of symptoms; 7-19 mild depression, 20-34 moderate depression, 35-60 indicate a severe depression.
MADRS total score (range 0-60) MADRS total score (range 0-60) change to BL/V0 (at V1) | baseline until end of titration phase at week 4 (V1)
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
ADHS-DC-Q total score (range 0-66) change to BL/V0 (V1) | baseline until end of titration phase at week 4 (V1)
  The ADHS-DC-Q consists of 18 items with a four-level response (not existing, slightly existing, moderately existing, strongly existing). The items ask about the current symptoms. The three scales are: lack of inattentiveness, hyperactivity and impulsiveness.
ADHS-DC-Q total score (range 0-66) change to BL/V0 (to V5) | baseline until end of treatment at week 16 (V5)
  The ADHS-DC-Q consists of 18 items with a four-level response (not existing, slightly existing, moderately existing, strongly existing). The items ask about the current symptoms. The three scales are: lack of inattentiveness, hyperactivity and impulsiveness.
QIDS-SR-16 total score (range 0-27) change to BL/V0 (V1) | from baseline to end of titration (week 4, V1)
  QIDS-SR-16 is a self-report measure of depression consisting of 16 items. Questions in the QIDS - SR-16 correlate with the nine DSM-IV symptom criterion domains, Including: Sleep disturbance (initial, middle, and late insomnia or hypersomnia), Sad mood, Decrease/increase in appetite/weight , Concentration , Self-criticism, Suicidal ideation, Interest, Energy/fatigue, Psychomotor agitation/retardation. Scoring is given from 0 to 3 whereas 0 indicates less impact, 3 highest impact in depression.
MADRS suicidal ideation score for all available visits | from enrollment to baseline (start of treatment, V0)
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on ten symptoms related to depression. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Reif, Prof. Dr. med., Study Chair — Department of Psychiatry, Psychosomatics and Psychotherapy University Hospital Frankfurt am Main - Goethe University
Locations (2):
- Germany (2):
  - Department of Psychiatry, Psychosomatics and Psychotherapy University Hospital Frankfurt am Main - Goethe University, Frankfurt
  - University Leipzig, Department of Psychiatry and Psychotherapy, Leipzig